CLINICAL TRIAL: NCT03944811
Title: Evaluation of Bone Height Gain Following Transcrestal Sinus Floor Elevation Using Piezoelectric Surgery Versus The Conventional Osteotome Technique in Patients With Atrophic Posterior Maxillae: A Randomized Controlled Clinical Trial
Brief Title: Bone Height Gain Following Transcrestal Sinus Floor Elevation Using Piezoelectric Surgery Versus The Conventional Osteotome Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Ashour, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 29011
Record Dates: First submitted 2019-05-07; First posted 2019-05-10 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcrestal sinus floor elevation using Summers technique (Active Comparator)
  Interventions: Procedure: Summers technique
- Transcrestal sinus floor elevation using piezoelectric surgery (Experimental)
  Interventions: Procedure: piezoelectric device

INTERVENTIONS:
Procedure: piezoelectric device — crestal approach will be used to augment the maxillary sinus with simultaneous implant placement
  Arms: Transcrestal sinus floor elevation using piezoelectric surgery
Procedure: Summers technique — Summers technique
  Arms: Transcrestal sinus floor elevation using Summers technique

SUMMARY:
Missing teeth usually result in functional and cosmetic deficits. Traditionally, they have been restored with dentures or fixed bridges. However, dental implants represent an excellent alternative which rely on the maintenance of a direct structural and functional connection between living bone and implant surface, which is termed osseointergration. When sufficient bone is available in maxilla, implant rehabilitation has shown high success rates of 84-92 %. Atrophy of the alveolar crest and pneumatization of the maxillary sinus limits the quality and quantity of residual bone, therefore complicating the placement of implants in the posterior maxillary area.

DETAILED DESCRIPTION:
Many solutions were suggested to overcome the problem of placing implants in the vertically compromised bone height in the maxillary posterior region. These solutions include the placement of short wide implants, long tilted zygomatic implants, vertical ridge augmentation and elevation of the sinus membrane to increase the available length for implant placement.

The use of short implants (<10 mm in length) is a reasonable solution that reduces the risk of interference with anatomic structures and claimed to have success rate as high as conventional implants. However, short implants have faced many challenges due to less bone-to-implant contact, more crestal bone resorption, and compromised crown-to-implant ratio. Another treatment option is the use of zygomatic implants. However, many complications may be associated with zygomatic implants such as oro-antral fistula formation, maxillary sinusitis, and peri-implant bleeding.

Vertical augmentation of the resorbed alveolar ridge is another treatment option. It can be done by onlay grafting, distraction osteogenesis and guided bone regeneration. Although success rates of various bone grafting techniques are high, there are many inherent disadvantages which include prolonged treatment times, raised treatment costs and increased surgical invasion associated with patient morbidity and potential complications.

To overcome these problems, elevation of the sinus membrane techniques were proposed, it can be performed either through a lateral window, or via a crestal access. The selection between these two techniques is mainly based on the remaining residual vertical subsinus bone height. Lateral approach of sinus elevation is indicated when the residual bone height is of 4 mm or less, while the crestal approach is used in case of residual ridge of 5-6 mm.

Many long term studies and systematic reviews have showed that osteotome mediated sinus floor elevation (OSFE) technique is a highly predictable method for rehabilitation of patients with atrophied posterior maxilla with survival rates ranging from 92 % to 100 %. However, endoscopic studies have demonstrated the risk of membrane perforation while performing transalveolar sinus floor elevation. Moreover, the Summers technique can cause some complications as headache and paroxysmal positional vertigo.

The piezoelectric internal sinus elevation (PISE) technique was first introduced by Sohn in 2009. Using piezoelectric ultrasonic vibration (25-30 kHz), the piezosurgery device cuts only mineralized structures precisely without cutting soft tissues even in case of accidental contact. Moreover, the cavitation effect produces a hydropneumatic pressure in the physiological saline solution that leads to atraumatic sinus membrane elevation. Another advantage of piezosurgery is its precision as the movement of the piezosurgery knife is very small, so the cutting precision is great and the patients discomfort is minimal. In addition, the air-water cavitation effect of the piezoelectric device sustains a blood-free surgical field which improves visualization of the surgical field. This technique overcomes the problem of benign paroxysmal positional vertigo caused by malleting during the osteotome mediated sinus floor elevation.

ELIGIBILITY:
Inclusion Criteria:

* • Patients having one missing upper posterior tooth residual bone height beneath maxillary sinus from 5-8 mm.

  * A minimum of 6 mm residual bone width at site of implant placement.
  * The recipient site of the implant should be free from any pathological conditions.
  * No diagnosed bone disease or medication known to affect bone metabolism.
  * Patients who are cooperative, motivated and hygiene conscious.
  * Patients having adequate inter-occlusal space of 8-10 mm.

Exclusion Criteria:

* Systemic conditions/diseases that contraindicate surgery.

  * Radiation therapy in the head and neck region or chemotherapy during the 12 months prior to surgery.
  * Patients who have any habits that might jeopardize the osseointegration process, such as current smokers.
  * Patients with parafunctional habits that produce overload on implant, such as bruxism and clenching.
  * Patients that have any pathology in the maxillary sinuses.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Amount of bone height gain | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Hassan El Barbary, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided